CLINICAL TRIAL: NCT03176680
Title: The Effects on Major Organ Complications on Esophagectomy of New Anesthetic ERAS (Enhanced Recovery After Surgery) Strategy: a Prospective Investigation
Brief Title: The Effects on Major Organ Complications on Esophagectomy of New Anesthetic ERAS Strategy: a Prospective Investigation
Acronym: ERAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201612093RINB
Record Dates: First submitted 2017-05-11; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Esophageal Cancer; Complication, Postoperative; Anesthesia
Keywords: Anesthesia,Esophagectomy,Esophageal cancer,Treatment outcome
MeSH Terms: conditions — Esophageal Neoplasms; Postoperative Complications

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluid therapy optimization (Experimental): Fluid loading to optimize stroke volume after induction.
  Interventions: Procedure: Fluid therapy optimization
- Fluid therapy normalization (No Intervention): No fluid loading after induction.

INTERVENTIONS:
Procedure: Fluid therapy optimization — colloid 250 mL bolus to increase stroke volume index (SVI). If the increase of SVI is more than 10% of baseline, repeat the bolus. If the increase of SVI is less than 10% of baseline, stop the bolus.
  Arms: Fluid therapy optimization

SUMMARY:
The goals of this study are to testify the effectiveness on enhancement recovery by new anesthetic ERAS (Enhanced recovery after surgery) strategy.

DETAILED DESCRIPTION:
ERAS (Enhanced recovery after surgery) strategy is extremely important for patients receiving esophagectomy including the preoperative preparation (smoking cessation, exercise prescription and nutrition prescription), intraoperative management, and postoperative analgesia and respiratory rehabilitation. However, despite the less invasive thoracoscopic esophagectomy and laparoscopic gastric tube reconstruction was developed, respiratory complications including acute lung injury (ALI) were observed up to 20% and associate with 50% of mortality. A new preventive anesthetic ERAS strategy including precise perioperative fluid management and preventive management after tracheal extubation should be developed.

Previous report indicated that none of the variables studied except fluid administration were shown as a risk factor for the development of respiratory complications on the multivariate analysis on esophageal surgery. However, there are rare prospective investigations of perioperative fluid administration strategy on postoperative complications after esophagectomy. Our group has studied on goal-directed fluid optimization and we found that the goal of optimization may differ for specific surgery. For esophagectomy, new anesthetic ERAS strategy should include precise preoptimized circulatory management and aggressive postoperative pulmonary care. Based on Frank-Starling law (stroke volume, SV, response to fluid therapy), a precise goal for perioperative goal-directed fluid therapy (GDFT) becomes possible in anesthetic practice. However, the effects of preoperative maximization of SV remain unknown. Following our study in last year, we planned to randomize 120 esophagectomy patients in the following 3 years into different GDFT groups (SV maximization and SV normalization groups). Postoperative THRIVE (Transnasal Humidified Rapid-Insufflation Ventilatory Exchange) therapy will be take place immediately after tracheal extubation. Blood samples will be obtained preoperatively to postoperative day 1 to measure lung injuries, kidney injuries as well as the inflammatory and oxidative markers. The clinical records will be collected (including extubation time, ICU stay, hospitalization days, 30-day mortality, 90-day mortality, readmission, postoperative cardiovascular, pulmonary, and renal complications, gastric tube related complications etc. ). The goals of this study are to testify the effectiveness on enhance recovery by new anesthetic ERAS strategy.

ELIGIBILITY:
Inclusion criteria:

* Patients with esophageal cancer
* Patients will undergo video-assisted thoracic surgical (VATS) esophagectomy and laparoscopic gastric tube reconstruction

Exclusion criteria:

* History of arrhythmia
* History of chronic obstructive pulmonary disease (COPD)
* With poor lung function test (FEV1 < 70% or FEV1/ forced vital capacity (FVC) < 70% of predicted)
* Preoperative creatinine more than 1.5 mg/dl

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-06-15 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | within 1 year after operation
  Length of ICU stay, total hospitalization days, 30-day mortality, 90-day mortality, postoperative pulmonary complications, cardiovascular complications, renal complications, prolonged extubation, readmission, gastric tube related complications

SECONDARY OUTCOMES:
Kidney injuries | Preoperative to postoperative day 1
  Elevated plasma creatinine
Lung injuries | Preoperative to postoperative day 1
  Change in the (PF ratio): ratio of arterial oxygen partial pressure (PaO2) to fractional inspired oxygen (FiO2)
Inflammatory markers | Preoperative to postoperative day 1
  Change in cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Jung Cheng, Principal Investigator — Anesthesiology Department, NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Test2, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided